CLINICAL TRIAL: NCT03305107
Title: The Effects of High-intensity Interval Exercise and Chocolate Milk on Glycemic Control and Cognitive Function in Children.
Brief Title: High-intensity Interval Exercise and Chocolate Milk on Blood Glucose and Cognition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Toronto Metropolitan University (Other)
Responsible Party: Principal Investigator, Nick Bellissimo, Study Director, Toronto Metropolitan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: REB2017- 088
Record Dates: First submitted 2017-09-29; First posted 2017-10-09 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Glycemic Response; Cognitive Function
Keywords: Child; Exercise; Chocolate milk; Blood glucose; Cognition; Appetite; Emotions; Cortisol
MeSH Terms: conditions — Motor Activity | interventions — Exercise; Water; Sitting Position

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exercise and Chocolate Milk (Experimental): Children will exercise on a cycle ergometer with a 3-min warm-up, 7 repeated bouts of 60-sec exercise at 90% of peak power output and 60-second recovery, and a 3-min cool down.
  Children will then drink 240mL of chocolate milk
  Interventions: Other: Exercise and Chocolate Milk
- Exercise and Water (Experimental): Children will exercise on a cycle ergometer with a 3-min warm-up, 7 repeated bouts of 60-sec exercise at 90% of peak power output and 60-second recovery, and a 3-min cool down.
  Children will then drink 240mL of water
  Interventions: Other: Exercise and Water
- Sitting and Chocolate Milk (Experimental): Children will quietly sit for 20 minutes Children will then drink 240mL of chocolate milk
  Interventions: Other: Sitting and Chocolate Milk
- Sitting and Water (Experimental): Children will quietly sit for 20 minutes Children will then drink 240mL of water
  Interventions: Other: Sitting and Water

INTERVENTIONS:
Other: Exercise and Chocolate Milk — High intensity interval exercise Chocolate Milk
  Arms: Exercise and Chocolate Milk
Other: Exercise and Water — High intensity interval exercise Water
  Arms: Exercise and Water
Other: Sitting and Chocolate Milk — Sitting Chocolate Milk
  Arms: Sitting and Chocolate Milk
Other: Sitting and Water — Sitting Water
  Arms: Sitting and Water

SUMMARY:
The purpose of this study is to determine the separate and combined effects of high-intensity interval exercise and chocolate milk on glycemic response, cognitive function, subjective appetite, and salivary cortisol among children aged 9-13 year old children.

DETAILED DESCRIPTION:
Twenty children 9-13 years of age will be recruited for this study. On four separate mornings, after a 10 hour overnight fast, each child will consume a standardized breakfast (including orange juice, a strawberry breakfast bar and a pear fruit cup) at home. Using a 2x2 factorial design, 2 hours after breakfast consumption, each participant will arrive in the lab (T=-20 min) and participate in high-intensity interval exercise or sit quietly for 20 min, followed by a treatment drink of chocolate milk or water (control) consumption in 10 min. During high-intensity interval exercise treatment, children will exercise on a cycle ergometer with a 3-min warm-up, 7 repeated bouts of 60-sec exercise at 90% of peak power output and 60-second recovery, and a 3-min cool down. Blood glucose will be measured via finger-prick at baseline (-20 min), 10, 30, 60, and 90 min. Cognitive functions will be measured using a battery of cognitive tests which assess verbal declarative memory, working memory, and executive functioning, and will be measured at baseline, 10. 30. 60, and 90 min. Subjective appetite and emotions will be measured using a 100-mm visual analogue scale (VAS) at baseline, 10, 30, 60, and 90 min. Salivary cortisol will be assessed from saliva samples collected using the passive drool method, and will be collected at baseline, 10 and 30 min.

ELIGIBILITY:
Inclusion Criteria:

* be between 9 and 13 years of age
* be healthy, and have been born at term
* not be taking any medications
* not have allergies to dairy or gluten.

Exclusion Criteria:

* Food sensitivities, allergies, or dietary restrictions
* Health, learning, emotional, or behavioural problems
* Receiving any medications
* Non-habitual breakfast eater (<5 days/week)

Ages: 9 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Actual)
Dates: Start 2017-07-08 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline Glycemic Response | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  Blood samples will be collected via finger-prick method to assess glycemic response (blood glucose, mmol/L)
Change from baseline verbal declarative memory | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  Cognitive function test of verbal declarative memory
Change from baseline working memory | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  The n-back test consists of 2 levels, 1-back and 2-back, where letters are presented on the screen one at a time. During the 1-back level, participants need to determine if the presented letter is the same as the one letter presented 1 before it or not (by selected 'match' or 'no match' on the side of the screen) and during 2-back need to do determine if it is the same letter as the one presented 2 letters prior.
Change from baseline executive functioning | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  The Stroop test consists of one word appearing on the screen written in either blue, red, yellow or green. There are 24 congruent trials where the presented word is the name of the colour it is written it (i.e. 'red' appearing in the colour red), 24 incongruent trials where the word written is a colour word different from the one it is written in (i.e. 'red' appearing in the colour green), and 10 neutral trials where non-colour words appear (i.e. 'tape' appearing in yellow). The participant is asked to tap the corresponding colour that the word is written in as quickly as possible.

SECONDARY OUTCOMES:
Change from baseline salivary cortisol response | baseline (-20 min), and 10 and 30 min post-drink consumption
  Saliva samples will be collected via passive drool method to assess salivary cortisol response (ug/dL)
Change form baseline Subjective Appetite | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  100-mm Visual Analogue Scales (VAS) will be used to assess appetite
Change from baseline aggression | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  100-mm Visual Analogue Scales (VAS) will be used to assess aggression
Change from baseline anger | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  100-mm Visual Analogue Scales (VAS) will be used to assess anger
Change from baseline excitement | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  100-mm Visual Analogue Scales (VAS) will be used to assess excitement
Change from baseline disappointment | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  100-mm Visual Analogue Scales (VAS) will be used to assess disappointment
Change from baseline happiness | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  100-mm Visual Analogue Scales (VAS) will be used to assess happiness
Change from baseline upset | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  100-mm Visual Analogue Scales (VAS) will be used to assess upset
Change form baseline frustration | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  100-mm Visual Analogue Scales (VAS) will be used to assess frustration
Change from baseline alertness | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  100-mm Visual Analogue Scales (VAS) will be used to assess alertness
Change from baseline sadness | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  100-mm Visual Analogue Scales (VAS) will be used to assess sadness
Change from baseline tension | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  100-mm Visual Analogue Scales (VAS) will be used to assess tension
Change from baseline exhaustion | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  100-mm Visual Analogue Scales (VAS) will be used to assess exhaustion
Change from baseline sleepiness | baseline (-20 min), and 10, 30, 60, and 90 min post-drink consumption
  100-mm Visual Analogue Scales (VAS) will be used to assess sleepiness

CONTACTS AND LOCATIONS:
Overall Officials: Nick Bellissimo, PHD, Study Director — School of Nutrition, Ryerson University
Locations (1):
- School of Nutrition, Ryerson University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kucab M, Bellissimo N, Prusky C, Brett NR, Totosy de Zepetnek JO. Effects of a high-intensity interval training session and chocolate milk on appetite and cognitive performance in youth aged 9-13 years. Eur J Clin Nutr. 2021 Jan;75(1):172-179. doi: 10.1038/s41430-020-00718-z. Epub 2020 Aug 19. PMID 32814852